CLINICAL TRIAL: NCT01242904
Title: Randomized Controlled Trial of Bimodal Solution for Peritoneal Dialysis: 24-Hour UF Efficiency Using Bimodal PD Solutions During the Long Dwell
Brief Title: Use of a Bimodal Solution for Peritoneal Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-10-460; 17193 (Other: Research Ethics Board)
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: End Stage Renal Disease
Keywords: dialysis solutions; renal replacement therapy; peritoneal dialysis; bimodal solution; glucose sparing therapy
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Icodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bimodal solution (Experimental): 200 mls of 30% glucose in sterile water is added by the patient to the usual icodextrin day dwell, to create the bimodal solution intraperitoneally
  Interventions: Drug: bimodal solution
- icodextrin (Active Comparator): 200 mls of icodextrin is added by the patient to the usual icodextrin day dwell
  Interventions: Drug: icodextrin

INTERVENTIONS:
Drug: bimodal solution — 200 mL of 30% glucose infused into the abdomen by the patient each morning for 6 weeks, added to the daytime dwell of approximately 2000 mL icodextrin that has been infused by the cycler
  Arms: bimodal solution
Drug: icodextrin — 200 mL of icodextrin infused into the abdomen by the patient each morning for 6 weeks, added to the daytime dwell of approximately 2000 mL icodextrin that has been infused by the cycler
  Arms: icodextrin

SUMMARY:
Peritoneal dialysis (PD) is the method of renal replacement therapy used by close to 200,000 end stage renal disease patients worldwide to help replace the functions that are no longer performed by their kidneys. An important advantage of PD is it offers an alternative to hemodialysis that can be safely performed by patients in their own homes. In PD, the peritoneal membrane that lines the abdomen acts as a dialyzer that allows the transfer of solutes and water between the membrane capillaries and a dialysis solution that is infused into the peritoneal cavity. PD dialysis solutions typically require high concentrations of glucose to adequately perform these functions. Over time the continued exposure of the peritoneal membrane to high concentrations of glucose can permanently damage the membrane. Icodextrin is a polyglucose molecule that has been developed for use in PD solutions that does not harm the peritoneal membrane. However, its use can lead to inadequate fluid removal. Recent research has focused on finding a PD solution, or combination of solutions, that will maximize the removal of toxic substances and metabolites while maintaining regulation of fluid and electrolyte balance in the body. A bimodal solution that combines glucose and icodextrin has been shown in observational studies to be effective and safe. The investigators propose a randomized, controlled, blinded study that will determine the effectiveness and safety of this bimodal fluid in a Canadian PD population. The investigators hypothesize that the use of the bimodal solution during the long (day) dwell will lead to an improvement in 24 hour ultrafiltration efficiency as compared to usual care using icodextrin for the long dwell.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide informed consent
2. Age greater than 18 years
3. Be stable Automated Peritoneal Dialysis (APD) patients for at least 6 weeks
4. Be APD patients who;

   1. Can be managed with an icodextrin long dwell AND
   2. Will use 4.25% and/or a 2.5% solution for at least one exchange overnight in at least 5 out of 7 days
5. Have residual urine volume <800 ml/24 hours
6. Long dwell must be or patient must tolerate at least an 8-10 hr long dwell.

Exclusion Criteria:

1. Scheduled Transplant in the next 1 year
2. Life expectancy < 3 mo (estimated by physician)
3. Participating in other trial that could influence outcome of this trial
4. Known icodextrin allergy
5. Currently using non-Baxter PD solutions
6. Systolic blood pressure < 90 mm Hg on more than three occasions during a seven day period, despite discontinuation of non-essential anti-hypertensives

Supplementary Exclusion Criteria (post Run-in phase):

1) Unsuccessfully completed 1 week run-in phase. Defined as:

1. Not using bimodal solution on 7 consecutive days during the run-in
2. Not tolerating the increased UF anticipated with the bimodal solution. Tolerating defined as:

i) Blood pressure drop below 90/50 on more than three occasions during a seven day period that cannot be corrected by reducing anti-hypertensives or other simple measures ii) Intolerable feeling of fullness with the bimodal solution iii) Allergic reaction (although all patients have already been exposed to icodextrin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-09-30 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2015-02-28 (Actual)

PRIMARY OUTCOMES:
net ultrafiltration efficiency in mL/g | Calculated at baseline and at the end of the 6 week intervention period
  Ultrafiltration Efficiency (UFE): UFE is defined as the amount of 24 hour net Ultrafiltration (UF) obtained for every gram of carbohydrate absorbed from the dialysis solution.
  1. 24-hour net ultrafiltration (in mL) is recorded automatically by the Automated Peritoneal Dialysis (APD) cycler.
  2. Carbohydrate absorption is determined by calculating the difference (in grams) between the amount of glucose (measured by lab analysis) in the 24 hr peritoneal effluent, and the amount of glucose in the patient's dialysis prescription.
  3. UFE will be calculated in mL/g (ie a divided by b)

SECONDARY OUTCOMES:
24-hour absolute total carbohydrate absorption | Calculated at baseline and at the end of the 6 week intervention period
  This will include both glucose and icodextrin absorption.
24-hour urine volume | Calculated at baseline and at the end of the 6 week intervention period
24-hour net sodium removal (in both peritoneal effluent and urine) | Calculated at baseline and at the end of the 6 week intervention period
Volume measures as calculated by bioimpedance analysis | Calculated at baseline and at the end of the 6 week intervention period
Weight | Calculated at baseline and at the end of the 6 week intervention period
  Used as an indicator of fluid retention
Mean and pulse arterial pressure | Calculated at baseline and at the end of the 6 week intervention period
Number of anti-hypertensive agents | Calculated at baseline and at the end of the 6 week intervention period
Renal (urine) solute clearance (Sodium, Urea, Creatinine) | Calculated at baseline and at the end of the 6 week intervention period
Peritoneal effluent solute clearance (Sodium, Urea, Creatinine) | Calculated at baseline and at the end of the 6 week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Arsh K Jain, MD, Principal Investigator — London Health Sciences Centre, Dept of Medicine, Victoria Campus, London Ontario
Locations (1):
- London Health Sciences Centre, South Street Hospital, Peritoneal Dialysis Unit, London, Ontario, Canada